CLINICAL TRIAL: NCT05965154
Title: Carrilizumab Combined With Bevacizumab Plus Capecitabine in a Second-line Prospective, One-arm Exploratory Study of Relapsed Metastatic Squamous Cell Carcinoma of Head and Neck
Brief Title: Calizumab Combined With Bevacizumab and Capecitabine in the Treatment of Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-LCYJ-ZF-09
Record Dates: First submitted 2023-04-23; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carrilizumab combined with bevacizumab plus capecitabine (Experimental): This study is a one-arm, exploratory study and does not involve randomization.There was only one trial group of carrilizumab plus bevacizumab plus capecitabine.
  Interventions: Drug: Carrilizumab, bevacizumab,capecitabine

INTERVENTIONS:
Drug: Carrilizumab, bevacizumab,capecitabine — 1. Carrilizumab: 200mg/ cycle, three weeks as a treatment cycle, the first day of each cycle, intravenous drip;
  2. Bevacizumab: 7.5mg/kg, intravenous infusion on the first day of each cycle, every 3 weeks for 1 cycle (Q3W);
  3. Capecitabine: 1250mg/m2, three weeks as a treatment cycle, oral twice a day (once in the morning and once in the evening; Stop the drug for 1 week after 2 weeks of treatment.

SUMMARY:
This is a prospective, one-arm exploratory second-line study of carrilizumab combined with bevacizumab plus capecitabine in relapsed metastatic squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, phase II clinical study. The study was intended to include histologically or cytologically determined squamous cell carcinoma of the head and neck, which the investigators assessed as metastatic. After the patients signed informed consent and met the screening criteria, the second-line patients received carrilizumab combined with bevacizumab and capecitabine until disease progression, intolerable toxicity, death, or the subject's decision to withdraw from the study for a maximum of two years.

Radiographic evaluations were performed using RECIST v1.1, and baseline evaluations were conducted within 28 days prior to enrollment. Tumor imaging evaluation was performed every 6 weeks (±3 days) from the first administration of the drug in the study. After reaching CR, patients entered the maintenance treatment period of carrilizumab. After 48 weeks, tumor imaging evaluation was performed every 12 weeks (±7 days). Imaging tests before signing the ICF, if within 28 days before starting treatment, can be used as screening tests.

During the study, participants will receive safety follow-up from the first dose of carrilizumab until 30 days after the last dose).

Experimental drugs: carrilizumab, bevacizumab, capecitabine

Administration regimen:

1. Carrilizumab: 200mg/ cycle, three weeks as a treatment cycle, the first day of each cycle, intravenous drip;
2. Bevacizumab: 7.5mg/kg, intravenous infusion on the first day of each cycle, every 3 weeks for 1 cycle (Q3W);
3. Capecitabine: 1250mg/m2, three weeks as a treatment cycle, oral twice a day (once in the morning and once in the evening; Stop the drug for 1 week after 2 weeks of treatment.

Duration of test plan and inclusion time:

1. Program selection time: 22 months.
2. Duration of the planned study: 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically determined, the investigators assessed patients with relapsed or metastatic squamous cell carcinoma of the head and neck. Including nasopharyngeal cancer, oral cancer, oropharyngeal cancer, hypopharyngeal cancer, laryngeal cancer, etc.
* The age range is between 18 and 85.
* Expected survival > 6 months.

Exclusion Criteria:

* Patients with uncured malignancies other than recurrent or metastatic squamous cell carcinoma of the head and neck diagnosed within 5 years prior to initial administration (excluding radical cutaneous basal cell carcinoma, cutaneous squamous epithelial carcinoma, and/or carcinoma in situ after radical excision).
* Previous treatment with anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that target another stimulus or synergistic inhibition of T cell receptors (e.g., CTLA-4, OX-40, CD137).
* Known allogeneic organ transplantation (except corneal transplantation) or allohematopoietic stem cell transplantation.
* other.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From the time a patient signs the ICF to the last dose, each patient will be followed up until death or withdrawal from the study or until 6 months after the last eligible patient is enrolled.
  Proportion of subjects assessed with CR or PR based on RECIST v1.1 criteria as a percentage of all enrolled patients

SECONDARY OUTCOMES:
Disease control rate | From the time a patient signs the ICF to the last dose, each patient will be followed up until death or withdrawal from the study or until 6 months after the last eligible patient is enrolled.
  Proportion of subjects assessed as CR, PR, or SD based on RECIST v1.1 criteria.
Progression-free survival time | From the time a patient signs the ICF to the last dose, each patient will be followed up until death or withdrawal from the study or until 6 months after the last eligible patient is enrolled.
  The time between the patient's first treatment date and any recorded tumor progression or death from any cause.
Overall survival time | From the time a patient signs the ICF to the last dose, each patient will be followed up until death or withdrawal from the study or until 6 months after the last eligible patient is enrolled.
  The time between the patient's date of first treatment and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jingqi Chen, MD, Study Chair — Principal Investigator

IPD SHARING:
Plan to Share IPD: No